CLINICAL TRIAL: NCT05857865
Title: Single-Session Psychotherapy for Young Kids Through Patient Engagement Techniques
Acronym: SPYKids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Specialized Services for Children and Youth (SCCY), Winnipeg, Manitoba (Unknown); Children's Hospital Research Institute of Manitoba (Other)
Responsible Party: Principal Investigator, Leslie E. Roos, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPYKids
Record Dates: First submitted 2023-03-31; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Mental Health Issue; Family Dynamics; Stress, Psychological; Stress, Emotional; Child Development
Keywords: single-session intervention; therapy; neurodevelopmental disorder
MeSH Terms: conditions — Stress, Psychological; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: The study will recruit caregivers with young children who have a neurodevelopmental disorder and who are currently on the waitlist for relevant services. Eligible caregivers (mothers, fathers, guardians) will be randomly assigned to either participate in one 90-minute single session intervention (SSI) in which a strategy will be developed to address a primary mental health concern or receive community family support services as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Caregivers in this group will participate in one 90-minute session delivered by a parenting coach via Zoom. This group will be asked to complete questionnaires at baseline, immediately post-program, approximately one month after the baseline assessment, and three months after the baseline assessment.
  Interventions: Behavioral: SPYKids
- Services as Usual (SAU) (Experimental): Caregivers in this group will not participate in a single-session intervention (SSI). Rather, this group will receive services as usual on the Specialized Services for Children and Youth (SCCY) waitlist. This group will be asked to complete questionnaires at baseline, approximately one month after the baseline assessment, and three months after the baseline assessment.
  Interventions: Other: Services as Usual (SAU)

INTERVENTIONS:
Behavioral: SPYKids — SSIs will be tailored to the parent areas of primary concern as identified in the pre-questionnaire. Participants will meet with the parent coach in a virtual 90-minute session to discuss coping strategies relevant to the identified concerns. Content will be informed by the baseline questionnaire and include psychoeducation with an explanation of 1 or 2 skills to manage a primary mental health issue (e.g., Emotion Regulation, Distress Tolerance, Communication), a brief practice of the skills (as appropriate), and an action plan for the family to apply the skills at home. Families will also be provided with recommendations for relevant services from our family-focused resource list. Please note, the session length may be extended to 120 minutes if an interpreter is required in order to provide equal opportunity for understanding the session content.
  Arms: Experimental
Other: Services as Usual (SAU) — Participants will receive links to the Manitoba 211 websites and a local organization's resource website with resources for adults and children. This resource is used to locate crisis, distress, and support phone lines, and counselling. Following completion of the 3-month survey, participants will receive a lab-developed comprehensive list of resources (also provided to participants in the SPYKids arm).
  Arms: Services as Usual (SAU)

SUMMARY:
The goal of this clinical trial is to compare outcomes between participants in the single-session psychotherapy for young kids (SPYKids) conditions and participants in the services as usual (SAU) condition. The main questions it aims to answer are:

* What is the feasibility and acceptability of SPYKids compared to services as usual?
* What are the changes in child mental health between the SPYKids group compared with the SAU group?

Participants will

* Fill out questionnaires at baseline, immediately post-program, approximately one month after the baseline assessment, and three months after the baseline assessment
* Meet with a parent coach in a virtual 90-minute session to discuss coping strategies relevant to their identified concerns

Researchers will compare participants in the SPYKids group with participants in the Services as Usual group to see if there are changes in child well-being, parent well-being, and parent self-efficacy.

DETAILED DESCRIPTION:
The coronavirus disease of 2019 (COVID-19) pandemic has contributed to elevated stress experienced by parents and caregivers of children with neurodevelopmental disorders (NDDs) resulting in increased demand for relevant specialized services. Current waitlists for NDD assessments following referral are approximately 12 months in Manitoba, with similar lengths of 6-30 months across Canada, which can result in children aging out of some early intervention services. The SPYKids program aims to provide families with help, encouragement, and motivation to cope with family stressors while on waitlists at local organizations through a single-session consultation model. A single-session intervention (SSI) is designed to increase parental ability to understand and address emergent mental health problems by teaching parents how to support children's emotional development and impulse control to reduce mental health problems, while reducing high-conflict parenting that can worsen mental health over time. The present study aims to test the feasibility and value of SSIs in a 2-arm randomized control trial which will include one 90-minute consultation with psychoeducation, identification of a primary mental health issue, an opportunity to practice the skills, and an action plan for the family to apply the skills independently. The long-term goal is to create an evidence-based accessible and rapidly deployable intervention to promote well-being for children with NDDs and their families.

ELIGIBILITY:
Inclusion Criteria:

* Manitoba resident with a Manitoba IP address
* Caregiver must be at least 18 years old
* Primary caregiver of 2-5-year-old child
* Must be on a waitlist for neurodevelopmental services in Manitoba

Exclusion Criteria:

* Living outside of Manitoba and/or internet protocol (IP) address outside of Manitoba
* Child is outside of the 2-5-year-old age range
* The caregiver is younger than 18 years old
* Not on a waitlist for neurodevelopmental services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Parent coach adherence to intervention protocol using the Fidelity Checklist | This measure is completed approximately 2 weeks after baseline. The first 6 items are completed by the parent coach at the end of the intervention and the last 23 items are completed immediately following the intervention (i.e., within a few minutes).
  29-item measure that assesses the extent to which the parent coach followed intervention protocols. Items are measured on a 5-point Likert scale with higher scores indicating greater adherence to protocols.
Feedback questionnaires pertaining to participant satisfaction with intervention protocol | The feedback questionnaires will be completed by participants immediately following the intervention (approximately 2 weeks after baseline).
  10-item questionnaire that measures parent satisfaction with intervention protocol. Participants respond to open-ended items regarding their satisfaction with the format of the SSI. This measure is qualitative in nature and no scores are generated.
Participant satisfaction with SSI format using the Program Feedback Scale | The Program Feedback Scale will be completed by participants immediately following the intervention (approximately 2 weeks after baseline).
  4-item questionnaire used to measure participant satisfaction with SSI. Participants respond to items on a 5-point Likert scale and are asked to rate the extent to which they feel the SSI will help with their identified problem. Higher scores indicate greater satisfaction.
Changes in child socioemotional and behavioural functioning between the SPYKids group compared with the SAU group - Strengths and Difficulties Questionnaire (SDQ) | The SDQ will be completed by participants at baseline, approximately 6 weeks from baseline (i.e., 1-month post-intervention for SPYKids group), and at 3 months post-intervention (approximately 12 weeks from baseline).
  A 25-item instrument developed to detect psychosocial problems in children aged 3-16 years. A value is given to each selection of "not true," somewhat true," and "certainly true." It measures five factors: emotional problems, conduct problems, hyperactivity/inattention problems, peer problems, and prosocial behaviour. All subscales include five items and range from 0-10. A total score can be summed from the first four factors; the total score ranges from 0-40, with higher scores indicating greater difficulties. Scores on the fifth factor of prosocial behaviour range from 0-10, with a lower score on this scale being less favourable.

SECONDARY OUTCOMES:
Changes in child socioemotional and behavioural functioning from pre- to 3- month post-intervention - Strengths and Difficulties Questionnaire (SDQ) | The SDQ will be completed by participants at baseline, approximately 1 month post-intervention and at 3 months post-intervention (approximately 12 weeks from baseline).
  A 25-item instrument developed to detect psychosocial problems in children aged 3-16 years. A value is given to each selection of "not true," somewhat true," and "certainly true." It measures five factors: emotional problems, conduct problems, hyperactivity/inattention problems, peer problems, and prosocial behaviour. All subscales include five items and range from 0-10. A total score can be summed from the first four factors; the total score ranges from 0-40, with higher scores indicating greater difficulties. Scores on the fifth factor of prosocial behaviour range from 0-10, with a lower score on this scale being less favourable.
Changes in parenting/caregiving stress from pre- to post-intervention - Parenting Stress Index (PSI; Short form) | The PSI will be completed by participants at baseline, approximately 1 month post-intervention and at 3 months post-intervention (approximately 12 weeks from baseline).
  A 36-item self-report measure completed by parents to measure stress level within the context of parenting. Participants respond to items on a 5-point Likert scale. Responses to each item in a sub-category are totalled to calculate three subcategory scores, which are summed to represent a total parenting stress score. Higher scores indicate higher levels of parenting stress. Normal scores fall within the 15th to 85th percentile, and scores above the 85th percentile represent clinically elevated levels of stress.
Changes in parental/caregiver depressive symptoms from pre- to post-intervention - Patient Health Questionnaire - 9 (PHQ-9) | The PHQ-9 will be completed by participants at baseline, approximately 1 month post-intervention and at 3 months post-intervention (approximately 12 weeks from baseline).
  A measure that assesses depressive symptoms using 8 items that align with diagnostic criteria with total possible scores ranging from 0 to 27, where higher scores are indicative of more severe symptoms.
Changes in parent anxiety symptoms -- Generalized Anxiety Disorder - 7 item scale (GAD-7) | The GAD-7 will be completed by participants at baseline, approximately 1 month post-intervention and at 3 months post-intervention (approximately 12 weeks from baseline).
  A brief self-report measure to screen for generalized anxiety disorder. Scores range from 0-21, with higher scores indicating more severe anxiety.
Changes in parent anger symptoms -- The Patient Records and Outcome Management Information System (PROMIS) Emotional Distress - Anger - Short-Form | The PROMIS-Anger will be completed by participants at baseline, approximately 1 month post-intervention and at 3 months post-intervention (approximately 12 weeks from baseline).
  A brief self-report measure used to assess the domain of anger. The items are measured on a 5-point Likert scale from "never" (1) to "always" (5). Total scores range from 5 to 25, with higher scores indicating more severe anger.

OTHER OUTCOMES:
Changes in parental/caregiver feelings of hope from pre- to post-intervention - Beck Hopelessness Scale - 4 (BHS) | The BHS will be completed by participants at baseline, approximately 1 month post-intervention and at 3 months post-intervention (approximately 12 weeks from baseline).
  A self-report measure that uses 20 true or false statements to assess feelings about the future, loss of motivation, and expectations. Higher total scores indicate greater hopelessness.
Changes in parental/caregiver perceived control/agency -- Perceived Control Single item (AGENCY) | The AGENCY will be completed by participants at baseline, immediately post-intervention (approximately 2 weeks after baseline), 1 month post-intervention, 3 months post-intervention (approximately 12 weeks from baseline).
  A single-item scale that measures perceived control of parents/caregivers by asking parents to rate their perceived sense of control on a scale from 1 to 10. Higher scores indicate less perceived control/agency.
Changes in parental/caregiver readiness to change - Readiness Ruler | The Readiness Ruler will be completed by participants at baseline, immediately post-intervention (approximately 2 weeks after baseline), 1 month post-intervention, 3 months post-intervention (approximately 12 weeks from baseline).
  A visual tool for parents/caregivers to rate the importance of making a change, their readiness to change, and confidence to change/take action on a 1-10 scale. Higher scores indicate ongoing attempts at changing.
Changes in parental/caregiver problem-solving strategies | The problem-solving strategies scale will be completed by participants immediately post-intervention (approximately 2 weeks after baseline), 1 month post-intervention, 3 months post-intervention (approximately 12 weeks from baseline).
  A measure that assesses the extent to which parents/caregivers are able to solve problems compared to pre-intervention on a 5-point scale from "much less able to solve problems" to "a lot more able to solve problems." Higher scores indicate more self-efficacy.
Changes in parental/caregiver perceived change in hopelessness | The perceived change in hopelessness scale will be completed by participants immediately post-intervention (approximately 2 weeks after baseline), 1 month post-intervention, 3 months post-intervention (approximately 12 weeks from baseline).
  A measure that assesses the extent to which parents/caregivers perceive changes in hopelessness compared to pre-intervention on a 5-point scale from "much more hopeless" to "a lot less hopeless." Higher scores indicate more hopefulness.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie E Roos, PhD, Principal Investigator — Assistant professor; Emily Cameron, PhD, Principal Investigator — Postdoctoral fellow
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (e.g. standardized questionnaire responses, aggregated program use data, sociodemographics linked to an identifier number) may be made available on public data platforms such as open science framework or a requirement by a granting agency or journal.
Supporting Information: Study Protocol
Time Frame: It would become available when the investigators publish the results of the study, approximately January 2024.
Access Criteria: Access will be based on the academic journal's level of access and requirements (e.g., subscription). Open access will be preferred at the time of journal selection, as possible, and preprint articles will be submitted online (e.g., psyarxiv.com) as possible based on journal requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT05857865/Prot_SAP_000.pdf